CLINICAL TRIAL: NCT04673682
Title: A Multicenter, Randomized, Single Blind, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety After Administration of CKD-845 in Males
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetic Profiles and Safety of CKD-845
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A106_01BE2011
Record Dates: First submitted 2020-11-06; First posted 2020-12-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Hypogonadism
Keywords: CKD-845
MeSH Terms: conditions — Hypogonadism | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 1. Treatment A: Reference drug(D309(Testosterone) 1 vial, once, i.m. inj.)
  2. Treatment B: Test drug(CKD-845(Testosterone) 1 vial, once, i.m. inj.)
  Interventions: Drug: D309; Drug: CKD-845
- Group 2 (Experimental): 1. Treatment B: Test drug(CKD-845(Testosterone) 1 vial, once, i.m. inj.)
  2. Treatment A: Reference drug(D309(Testosterone) 1 vial, once, i.m. inj.)
  Interventions: Drug: D309; Drug: CKD-845

INTERVENTIONS:
Drug: D309 — D309(Testosterone) 1 vial, Once, IM injection
  Other Names: Reference Drug
Drug: CKD-845 — CKD-845(Testosterone) 1 vial, Once, IM injection
  Other Names: Test Drug

SUMMARY:
A clinical trial to evaluate the pharmacokinetic profiles and safety of CKD-845.

DETAILED DESCRIPTION:
A phase 1 clinical trial to evaluate pharmacokinetics and safety in male after administration of CKD-845 and D309.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Male over 19 years old and under 65 years old at screening.
2. Serum total testosterone level under 3.0 ng/mL at screening.
3. Subjects who had 18.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5 kg/m2 and a total body weight ≥ 55 kg.

   * Body Mass Index(BMI) = Weight(kg) / [Height(m)]2
4. Subjects without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years, except for hypogonadism.
5. Subjects who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, vital signs, ECG etc.).
6. Subjects who voluntarily signed an informed consent form approved by the Institutional Review Board(IRB) of each clinical study site and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content of the clinical trial.
7. Subjects who consent to the use of reliable contraception during the clinical trial. Subjects who have no plan of pregnancy and agree to not donate his sperm during the study period and up until 180 days after the last administration of investigational product.
8. Subjects with the ability and willingness to participate during the study period.

Exclusion Criteria:

1. Subjects with a medical evidence or a history (excluding a hypogonadism, dental history of periodontal surgery, impacted wisdom teeth removal, etc.) of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune disease.

   1-1. Subjects with a severe acute/chronic physical and mental conditions that can increase risk or interfere with the interpretation of the results of test.

   1-2. Subjects who have a androgen-dependent tumor(e.g., prostate cancer, male breast cancer).

   1-3. Subjects with hypercalcemia associated with malignant tumors.

   1-4. Subjects with or with a history of liver tumors.

   1-5. Subjects with bone metastasis of cancer.

   1-6. Subjects being treated for an enlarged prostate.

   1-7. Subjects who have severe alcohol and/or drug abuse history within a year from screening.

   1-8. Insulin-dependent diabetes mellitus or uncontrolled non-insulin- dependent diabetes mellitus.
2. Subjects with the following laboratory test results at screening:

   2-1. AST, ALT exceeding 2.5 times from the upper limit of normal.

   2-2. Total bilirubin exceeding 2.5 times from the upper limit of normal.

   2-3. Subjects had renal impairment(eGFR < 60 mL/min/1.73 m2)

   2-4. Positive results of virus/bacterial test and/or urine drug test at screening.

   2-5. Systolic blood pressure >150 mmHg or <90 mmHg and/or diastolic blood pressure >60 mmHg or >95 mmHg at sitting position.
3. History of regular alcohol consumption exceeding 210 g/week within 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g, 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL of wine (12%) = 12 g).
4. Subjects who smoked more than 20 cigarettes per day within 6 months prior to screening.
5. Subjects who had been administered investigational product(s) from other clinical study or bioequivalence study within 180 days prior to the first dose of this study(except when subject have not taken investigational product(s)).
6. Subjects who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first dose of investigational product(s).
7. Subjects who had taken any contraindication drug(s)(Drug influencing the level of serum testosterone, modulating activity of testosterone and which have drug interaction) within 28 days prior to the first dose of investigational product(s).
8. Subjects who use of oral anticoagulants (with the exception of low-dose aspirin) within 28 days prior to the first dose of investigational product(s).
9. Subjects who use the testosterone pellet within 90 days prior to the first dose of investigational product(s).
10. Subjects who use of any injectable testosterone preparations within 28 days prior to the first dose of investigational product(s).
11. Subjects who use oral testosterone products within 7 days prior to the first dose of investigational product(s).
12. Subjects who use of supplements (e.g., saw palmetto, phytoestrogen, androstenedione, DHEA, niacin, fish oil etc.) prior to the first dose of investigational product(s).
13. Subjects who have hypersensitivity of investigational products and its components.
14. Subjects who donated whole blood within 60 days or blood components within 30 days prior to the first dose of the investigational product(s).
15. Subjects who were deemed inappropriate to participate in the study by the investigator.

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 47 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Baseline corrected AUCt of CKD-845 | up to 70 days
  AUCt: Area under the concentration-time curve from time zero to time
Baseline corrected Cmax of CKD-845 | up to 70 days
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
Baseline corrected AUCinf of CKD-845 | up to 70 days
  AUCinf: Area under the concentration-time curve from zero up to infinity
Baseline corrected Tmax of CKD-845 | up to 70 days
  Tmax: Time to maximum plasma concentration
Baseline corrected t1/2 of CKD-845 | up to 70 days
  t1/2: Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, M.D., PhD., Principal Investigator — Jeonbuk University Hospital; An-Hye Kim, M.D., PhD., Principal Investigator — CHA Bundang Medical Center; Hyewon Chung, M.D., PhD., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Jeonbuk University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No